CLINICAL TRIAL: NCT03544424
Title: A Study of Physical Activity paTTerns and Major Health Events in Older People With Implantable Cardiac Devices
Acronym: PATTErn
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Joanne Taylor, Clinical Fellow in Cardiology, Postgraduate Student, University of Manchester
Other Study IDs: 215964
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity; Aging; Cardiac Disease
MeSH Terms: conditions — Motor Activity; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: People over 60 years of age with a Medtronic CareLink® compatible CIED in situ recruited from the Manchester University NHS Foundation Trust, England, UK
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
An observational study of physical activity patterns in 150 older adults with cardiac implantable electronic devices (CIED)

DETAILED DESCRIPTION:
Study Type: observational, investigator led Study Design: observational model: cohort (retrospective) Population: 150 people over 60 years of age with a Medtronic CareLink® compatible CIED in situ recruited from the Manchester University NHS Foundation Trust, England, UK Data collection: daily PA measures, demographic details, co-morbidity status, physical frailty assessment, functional status, quality of life (QOL) and NEHA data Consent: for participation in the study, physical frailty assessment, additional collection of retrospective CIED data, and access to electronic patient records Data sources: CIED downloads, self-report questionnaire, physical measurements (height, weight, hand grip strength, gait speed), electronic hospital records, HES (hospital episode statistics) data Results analysis: data will be analysed to investigate: daily PA variability; the association between PA and NEHAs, and the impact of frailty on PA patterns

ELIGIBILITY:
Inclusion Criteria:

1. Age 60+ years
2. Functioning CIED in situ for at least 6 months
3. Medtronic manufactured device compatible with CareLink® Cardiac Compass application (platform which measures and stores physiological parameters)
4. Lives in the Greater Manchester area
5. Able and willing to given written, informed consent to enter the study

Exclusion Criteria:

1. Faulty or incompatible device
2. Immobile (unable to walk in upright position)
3. Active participant in a clinical trial which does not allow concurrent recruitment into this study
4. People unable to consent in the English language (including the understanding of study literature which is published in English only)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People 60 years or older with CIED in situ for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Greenstein, MBChB, PhD, Study Director — Manchester University
Locations (1):
- Manchester Heart Centre, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Cohort
Started | 183
Completed | 183
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Cohort
Number analyzed (Participants) | 183
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [72 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 183
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 183

OUTCOME MEASURES:

1. Primary Outcome: Non-elective Hospital Admissions
Description: Non-elective hospital admissions, as defined as an emergency admission to an National Health Service (NHS) hospital within England or Wales for any reason. Data collected from NHS England.
  Number of Participants With Non-elective Hospital Admissions.
Time Frame: Retrospective: 12 months prior to enrolment (retrospective data spans 12 months prior to enrolment)
Population: People over 60 years with compatible implanted cardiac device
Measure: Count of Participants; unit: Participants
Groups:
- Low Activity: Participants with mean physical activity <1 hour per day
- Medium/High Activity: Participants with mean physical activity >1 hour per day
Arm/Group | Low Activity | Medium/High Activity
Number analyzed (Participants) | 33 | 107
Participants
  Non-elective hospitalisation | 2 | 3
  No non-elective hospitalisation | 31 | 104

2. Secondary Outcome: Frailty
Description: Frailty as per Fried criteria
  Fried frailty criteria is a score between 1-5. A score of 0-1 = not frail A score of 2 = pre-frail A score of 3+ = frailty
  Reference:
  Fried, L. P., Tangen, C. M., Walston, J., Newman, A. B., Hirsch, C., Gottdiener, J., ... & McBurnie, M. A. (2001). Frailty in older adults: evidence for a phenotype. The journals of gerontology series a: biological sciences and medical sciences, 56(3), M146-M157.
Time Frame: 30 days
Population: 140 participants had adequate activity data from devices
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 140
Participants
  Frailty | 16
  Pre-frailty | 74
  Not frail | 50

ADVERSE EVENTS:
Time Frame: 1 day
Description: No prospective follow-up
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/183
Serious Adverse Events (participants affected / at risk) | 0/183
Other Adverse Events (participants affected / at risk) | 0/183

LIMITATIONS AND CAVEATS:
This was a cross-sectional study. Recruitment was limited due to COVID-19, therefore study design was adapted. The primary outcome was non-elective hospital admissions, however there were too few events to facilitate the primary analysis. Secondary outcome of the study was to investigate the association between physical activity as measured by cardiac device and frailty.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03544424/Prot_SAP_000.pdf